CLINICAL TRIAL: NCT04528017
Title: Clinical Comparison of 2 Daily Disposable Contact Lenses - Pilot Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-P004
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-09

CONDITIONS: Refractive Errors; Myopia
Keywords: Daily disposable contact lenses
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PRECISION1, then Clariti 1-Day (Other): Verofilcon A contact lenses worn first, with somofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Somofilcon A contact lenses
- Clariti 1-Day, then PRECISION1 (Other): Somofilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Somofilcon A contact lenses

INTERVENTIONS:
Device: Verofilcon A contact lenses — Spherical soft contact lenses for daily disposable wear
  Other Names: PRECISION1™
Device: Somofilcon A contact lenses — Spherical soft contact lenses for daily disposable wear
  Other Names: CooperVision® clariti® 1 day; Clariti 1-Day

SUMMARY:
The primary objective of this study is to evaluate the overall performance of PRECISION1 contact lenses when compared to Clariti 1-Day contact lenses.

DETAILED DESCRIPTION:
Subjects are expected to attend 3 study visits and wear the PRECISION1 and Clariti 1-Day study lenses in a crossover design for approximately 8 days of exposure to each study lens type. The expected duration of subject participation is up to 22 days.

ELIGIBILITY:
Key Inclusion Criteria

* Subject must be able to understand and must sign an Institution Review Board (IRB) approved Informed Consent Form.
* Successful wear of soft contact lenses in both eyes for a minimum of 5 days per week and 10 hours per day during the past 3 months.
* Willing to wear contact lenses for at least 16 hours per day on one of the days with each lens type.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any ocular condition that contraindicates contact lens wear.
* Previous or current habitual wearer of PRECISION1, Clariti 1-Day, or DAILIES TOTAL1 contact lenses.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Project Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (4):
- United States (4):
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6402, Medina, Minnesota
  - Alcon Investigator 6313, Powell, Ohio
  - Alcon Investigator 8028, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 investigative sites located in the United States.
Pre-assignment Details: Of the 56 subjects enrolled in the study, 1 subject was discontinued prior to randomization. This reporting group includes all randomized subjects as treated (55).
Units Other Than Participants: eyes
Groups:
- PRECISION1, Then Clariti 1-Day: Verofilcon A contact lenses worn first, with somofilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
- Clariti 1-Day, Then PRECISION1: Somofilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
Period: First Wear Period (8 -0/+3 Days)
Arm/Group | PRECISION1, Then Clariti 1-Day | Clariti 1-Day, Then PRECISION1
Started | 27; 54 eyes | 28; 56 eyes
Completed | 27; 54 eyes | 28; 56 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: Second Wear Period (8 -0/+3 Days)
Arm/Group | PRECISION1, Then Clariti 1-Day | Clariti 1-Day, Then PRECISION1
Started | 27; 54 eyes | 28; 56 eyes
Completed | 27; 54 eyes | 28; 56 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | PRECISION1, Then Clariti 1-Day | Clariti 1-Day, Then PRECISION1 | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (7.7) | 33.3 (7.5) | 33.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) With Study Lenses
Description: Distance VA was assessed with study lenses in place. VA was collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity. No formal hypothesis was predefined for the primary endpoint. No inferential testing was performed.
Time Frame: Day 8 (-0/+3 days) after 10 (-2/+6) hours of wear, each study lens type
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- PRECISION1: Verofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -0/+3 days in a daily disposable modality
- Clariti 1-Day: Somofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -0/+3 days in a daily disposable modality
Arm/Group | PRECISION1 | Clariti 1-Day
Number analyzed (Participants) | 55 | 55
Number analyzed (eyes) | 110 | 110
logMAR | -0.13 (0.07) | -0.15 (0.06)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, up to 22 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- PRECISION1 Ocular; PRECISION1 Nonocular: Events reported in this group occurred while exposed to the verofilcon A contact lenses
- Clariti 1-Day Ocular; Clariti 1-Day Nonocular: Events reported in this group occurred while exposed to the somofilcon A contact lenses
Arm/Group | Pretreatment | PRECISION1 Ocular | PRECISION1 Nonocular | Clariti 1-Day Ocular | Clariti 1-Day Nonocular
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/110 | 0/55 | 0/110 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/110 | 0/55 | 0/110 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/110 | 0/55 | 0/110 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT04528017/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT04528017/SAP_001.pdf